CLINICAL TRIAL: NCT06779604
Title: Comparison of the Anesthetic Effects of Dexmedetomidine and Dexamethasone Added as Adjuvant to Ultrasonography-Guided Infraclavicular Brachial Plexus Block in Upper Limb Surgery
Brief Title: Dexmedetomidine and Dexamethasone Added as Adjuvant Infraclavicular Brachial Plexus Block in Upper Limb Surgery
Status: Recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Head of Anesthesia and reanimation, Umraniye Education and Research Hospital
Other Study IDs: UERH-AR-ZT-11
Record Dates: First submitted 2024-12-22; First posted 2025-01-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain; Anesthesia; Acute Pain
Keywords: infraclavicular nerve block; dexmetomidine; dexamethosone
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Dexmedetomidine: (n:22): A total volume of 30 mL of 0.5% bupivacaine, 14 mL of 2% lidocaine and 50 μgr of dexmedetomidine in 1 mL of normal saline is administered to the patients.
  Interventions: Procedure: Infraclavicular Block with Dexmedetomidine and Dexamethasone
- GroupDexamethasone: (n:22): Patients are administered 0.5% bupivacaine 15 mL, 2% lidocaine 14 mL and 4 mg dexamethasone in 1 ml normal saline with a total volume of 30 mL
  Interventions: Procedure: Infraclavicular Block with Dexmedetomidine and Dexamethasone

INTERVENTIONS:
Procedure: Infraclavicular Block with Dexmedetomidine and Dexamethasone — Infraclavicular block with Dexmedetomidine and Dexamethasone was performed at least 30 min before the start of the operation. The patient was positioned in a supine position arms at the sides or in 90 degree abduction, head turned to the other side. Infraclavicular block was performed with the lateral sagittal technique, while the USG probe was placed under the clavicle and medial to the coracoid process, providing a brachial plexus image in the form of a hyperechoic outer ring and hypoechoic circles, like a classic honeycomb image. A local anesthetic mixture was injected with a 100 mm block needle with negative aspiration and its spread in tissue planes was observed.
  If the VAS score was 3 or above, tramadol 1 mg kg-1 was administered as an analgesic drug.

SUMMARY:
The aim of this study was to investigate the effect of dexmedetomidine and dexamethasone added during USG-guided infraclavicular block on block onset time, total block time and time to first analgesic need in patients undergoing upper extremity surgery.

DETAILED DESCRIPTION:
Brachial plexus blocks are successfully applied for perioperative/postoperative analgesia in upper extremity surgical procedures. These blocks include infraclavicular, supraclavicular, interscalene, and axillary blocks. The reason why infraclavicular block is preferred is that it provides comprehensive anesthesia/analgesia of the upper extremity. While the axillary approach may fail to block the musculocutaneous nerve that causes tourniquet pain, the interscalene and supraclavicular approaches generally fail to provide anesthesia in the distribution of the ulnar nerve. Other advantages include the lower risk of lung and pleural puncture compared to interscalene and supraclavicular blocks and the lower probability of injury to neurovascular structures due to the location of the block, unlike the interscalene approach.

Local anesthetics are used to block conduction in nerve fibers during brachial plexus blocks. Studies have shown that the commonly used bupivacaine and ropivacaine 0.25% concentrations are not recommended for anesthesia. Bupivacaine 0.5% and ropivacaine 0.5% have been shown to be similar in terms of sensory and motor block onset time, total sensory and motor block duration, analgesia duration, anesthesia duration, paresis and paralysis incidence. The minimum dose of bupivacaine 0.5% required for complete sensory block was determined as 14mL, but the onset time of the block performed at this low dose was recorded as a late onset of 40 minutes (30-45 minutes). It was observed that the onset time decreased to as short as 15 minutes (min) after the application of 30mL bupivacaine 0.5%. In order to reduce the amount of local anesthetic used, to avoid local anesthetic toxicity, to shorten the block onset time and to extend the postoperative analgesia period, a different local anesthetic or adjuvants were used together with bupivacaine. Bupivacaine used with lidocaine has been observed to have a faster onset of action. Other adjuvants added to accelerate the onset of block and improve the quality of the block include alpha-2 agonists (clonidine and dexmedetomidine), opioids (fentanyl and tramadol), and steroids (dexamethasone). Dexmedetomidine is an adjuvant that is an alpha-2 adrenergic agonist and has been observed to have a synergistic effect with local anesthetics and to prolong their duration of activity. The addition of dexmedetomidine 50 µg and 75 µg has been associated with a decrease in the time to onset of sensory and motor block, a decrease in postoperative morphine consumption, and an increase in the duration of sensory block, motor block, and the time to first morphine request. Dexmedetomidine 75 µg has been associated with an increased incidence of preoperative and intraoperative hypotension episodes. Dexamethasone, a perineural adjuvant, has been shown in many studies to significantly shorten the onset of sensory and motor block and prolong the duration of analgesia. Perineural dexamethasone is more commonly used intravenously for block. Currently, many studies have compared the effects of various perineural dexamethasone doses, such as 1 mg, 2 mg, 4 mg, 5 mg and 8 mg, on block, but the results remain controversial. Studies have shown that there is no difference in safety and efficacy between 4 and 8 mg perineural dexamethasone. Another study reported that 4 mg perineural dexamethasone constitutes a ceiling dose for prolonging the duration of analgesia when used with local anesthetics for block.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* ASA I-II

Exclusion Criteria:

* Under 18 years of age and older than 70 years of age,
* presence of brachial plexus injury,
* patients with bleeding diathesis,
* presence of allergy, -contralateral diaphragmatic paralysis, -
* presence of nerve injury secondary to trauma,
* pre-existing neuropathy of the surgical extremity,
* presence of severe pulmonary,
* renal and hepatic disease,
* congestive heart failure (NYHA stage 3-4),
* uncontrolled diabetes mellitus,
* history of neuromuscular disease,
* patients with extreme obesity or malnutrition (BMI > 30 kg-1m2 or BMI <20 kg-1m2),
* presence of epilepsy,
* history of peripheral vascular disease,
* history of chronic pain or fibromyalgia,
* pregnant and lactating patients,
* patients with local infection at the injection site,
* patients undergoing general anesthesia due to inadequacy of the block,
* patients refusing to give informed consent,
* history of recreational substance use, and chronic narcotic-based painkillers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 44 adult patients 18 to 70 years, American Society of Anesthesiologists (ASA) I-II who underwent upper extremity surgery were included in Orthopedics and Traumatology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
infraclavicular block onset time | 24 -48 hours
  Sensory block / motor block onset time
postoperative analgesic drug requirement | 24 -48 hours
  opioid total amount micrograms
infraclavicular total block time | 24 -48 hours
  block time hours

SECONDARY OUTCOMES:
investigate the effects on VAS score and sedation level in the first 24 hours postoperatively | 24 -48 hours
  VAS score
advers event Perioperative and postoperative period | 24 -48 hours
  Nausea,Vomiting,Hypotension,Bradycardia, Nerve damage

CONTACTS AND LOCATIONS:
Overall Officials: ZELİHA TUNCEL, ASC PROF, Study Director — Umraniye ERH
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No